CLINICAL TRIAL: NCT05723042
Title: Effects of Neuromuscular Electrical Stimulation With and Without Constraint Induced Movement Therapy on Upper Limb Function in Children With Erb's Palsy
Brief Title: Neuromuscular Electrical Stimulation With and Without Constraint Induced Movement Therapy in Erb's Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REC/RCR & AHS/22/0749
Record Dates: First submitted 2023-01-24; First posted 2023-02-10 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: Erb's Palsy
MeSH Terms: conditions — Brachial Plexus Neuropathies

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EMS with CIMT group (Experimental)
  Interventions: Other: EMS with CIMT
- EMS Group (Active Comparator)
  Interventions: Other: EMS

INTERVENTIONS:
Other: EMS with CIMT — The interventions are consisted of 3weeks of casting the unaffected limb followed by 5 weeks of transference activities.The assisting hand assessment AHA was used to measure bimanual activity performance at baseline,8 weeks, 16 weeks. 20-minute application of currents and resistance exercises for the respective muscles of the area. The intervention group with 11 patients underwent a program of CIMT for one hour daily for 14 consecutive days or two hours per day, six days per week and a total of 12 weeks. A follow-up will be performed 12 weeks after the intervention. The healthy upper limb will be immobilized by orthosis or cast for six hours a day . Electrotherapy will be applied with TENS for 15 minutes at intervals of 1000ms and with a pulse duration of 50ms. The square wave will be chosen to ensure that there will be sufficient muscle contraction
  Arms: EMS with CIMT group
Other: EMS — this group will only receive baseline exercises (ROM and flexibility exercises) than apply electrical stimulations at specific motor points. Electrotherapy will be applied with TENS for 15 minutes at intervals of 1000ms and with a pulse duration of 50ms. The square wave will be chosen to ensure that there will be sufficient muscle contraction
  Arms: EMS Group

SUMMARY:
Erb's Duchenne paralysis constitutes the single commonest form of brachial plexus injury, brachial plexus injury (BPI) is unfortunately a rather common injury in newborn children. Incidence varies between 0.15 and 3 per 1000 live births in various series and countries. The constraint-induced movement therapy (CIMT) has been used to promote functional gains in individuals with neurological dysfunctions .The constraint-induced movement therapy consists of constraining movement of the non-affected upper extremity and providing intensive training to the involved upper extremity. Neuromuscular electrical stimulation (NMES) has been used for muscle strengthening, maintenance of muscle mass and strength during prolonged periods of immobilisation, selective muscle retraining, and the control of oedema.The aim of this study is to compare the effects of Neuromuscular Electrical Stimulation with and without Constraint Induced Movement Therapy on Upper limb Function in Children with Erb's Palsy.

It is a Randomized Controlled Trial.The sample size calculated by using OpenEpi or GPower. Data will be collected from Jinnah Hospital,Children Hospital,Lahore medical city hospital,Farooq hospital,Rising sun institute and PSRD. The patients will be selected through non-probability convenience sampling,will be divided into two groups. The Group A will receive habituation exercises for six weeks, three times per week for thirty minutes, along with application of neuromuscular electrical stimulation for a period of 6 weeks four times a week and perform Constrained induced movement therapy techniques, each for 8 weeks.The interventions are consisted of 3weeks of casting the unaffected limb followed by 5 weeks of transference activities.. The Group B will be given neuromuscular electrical stimulation for a period of 6 weeks four times a week.Range of motion ,Flexibility exercises will be given as baseline treatment to both groups. The arm function was evaluated by the Mallet score system, while active abduction and external rotation range of motion were measured by a standard universal goniometer. Data will be analyzed by SPSS 25.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 2.5 to 8 years years
* Clinically diagnosed with erb's palsy/brachial plexus palsy
* Ability to cooperate with assessments and therapy
* Full passive ROMs in all motions at the shoulder, elbow, and wrist joints

Exclusion Criteria:

* Cognitive impairment
* Contracture in the affected upper extremity
* Injured unaffected arm
* Visual problems likely to interfere with treatment/testing
* Previous orthopedic or neurological surgery
* Previous application of CIMT

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 22 (Actual)
Dates: Start 2023-01-13 (Actual); Primary Completion 2023-03-01 (Actual); Study Completion 2023-03-28 (Actual)

PRIMARY OUTCOMES:
Change in Mallet scale Scores | Baseline, 8th week and 16th week
  The Mallet grading remains the most commonly used system in several obstetric brachial plexus centers. One feature of the Mallet score is that each grade is translated into certain degrees of deficiencies in both shoulder abduction and external rotation.
Change in Box and block test scores | Baseline, 8th week and 16th week
  the BBT has been commonly used in the pediatric field. It is particularly suitable for children for several reasons. First, the evaluation method of the BBT examines essential components of manual dexterity for developing children, such as grasping, holdi

CONTACTS AND LOCATIONS:
Overall Officials: Muneeb Iqbal, PhD, Principal Investigator — Riphah International University
Locations (1):
- Jinnah Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gonçalves RV, Araujo RCd, Ferreira VKG. Effect of reaching training combined with electrical stimulation in infants with brachial plexus palsy: a single subject design. Fisioterapia e Pesquisa. 2021;28:32-8.
- [Background] Justice D, Awori J, Carlson S, Chang KW, Yang LJ. Use of neuromuscular electrical stimulation in the treatment of neonatal brachial plexus palsy: A literature review. The Open Journal of Occupational Therapy. 2018;6(3):10
- [Background] Sakzewski L, Ziviani J, Boyd R. Systematic review and meta-analysis of therapeutic management of upper-limb dysfunction in children with congenital hemiplegia. Pediatrics. 2009 Jun;123(6):e1111-22. doi: 10.1542/peds.2008-3335. Epub 2009 May 18. PMID 19451190